CLINICAL TRIAL: NCT01918462
Title: Protective Immune Mechanisms in Alcoholic Hepatitis
Acronym: AHIL
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: AHIL; AUH (Other: Aarhus University hospital)
Record Dates: First submitted 2013-06-25; First posted 2013-08-07 (Estimated); Last update posted 2021-04-29 (Actual); Status verified 2018-10

CONDITIONS: Alcoholic Hepatitis
Keywords: Alcoholic hepatitis; IL-22; Kupffer cells
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma, PBMC's, hepatic leukocytes
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Alcoholic hepatitis: Patients with alcoholic hepatic; cases.
- Healthy controls: Persons undergoing hepatic resection; controls.

SUMMARY:
The purpose of this study is to investigate the production, effects and interactions of the hepato-protective cytokine interleukine (IL)-22 in patients with alcoholic hepatitis.

DETAILED DESCRIPTION:
The investigators will study hepatic biopsies from patients with alcoholic hepatitis. In these biopsies, the investigators will assess the production of IL-22 and which cells produce the cytokine. The investigators will study the expression of the IL-22 receptor and also the production of the IL-22 binding protein, which can inhibit the actions of the cytokine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of alcoholic hepatitis:
* relevant history of alcohol consumption (>40g/day for a minimum of 6 months with cessation of consumption no earlier than 3 months prior to admission)
* bilirubin > 80 mol/l
* neutrophil granulocytes > 10x10^9/L
* exclusion of other liver pathology including biliary disease
* histological verification on liver biopsy
* Written, informed consent

Exclusion Criteria:

* Other chronic inflammatory or autoimmune diseases
* Severe, acute bacterial infection (peritonitis, sepsis, pneumonia, urinary tract infection etc.)
* Cancer
* Prednisolon or pentoxifylline treatment within the past 8 weeks
* Pregnancy

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Department of hepatology and gastroenterology V, Aarhus University hospital
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-04-20 (Actual)

PRIMARY OUTCOMES:
Frequency of IL-22-producing cells | at day 1 ( the day of diagnosis/arrival to the department)
  This will be detected in hepatic biopsies taken at inclusion to the study.

SECONDARY OUTCOMES:
IL-22 binding protein | at day 1 ( the day of diagnosis/arrival to the department)
  This will be detected in hepatic biopsies taken at inclusion to the study.
IL-22 receptor | at day 1 ( the day of diagnosis/arrival to the department)
  This will be detected in hepatic biopsies taken at inclusion to the study.
Signalling molecules and markers of hepatocyte destruction | at day 1, at day 7 and at day 90 after diagnosis.
  Thse measurements will be done on blood samples drawn at inclusion, at day 7 and at day 90 after diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Sidsel Støy, Phd student, Principal Investigator — Department of hepatology and gastroenterology, Aarhus University Hospital
Locations (1):
- Department of Hepatology and gastroenterology V, Aarhus university hospital, Aarhus, Denmark